CLINICAL TRIAL: NCT00972426
Title: A Randomized, Parallel, Open-label Study to Evaluate Efficacy and Safety Effects Using Mikelan® LA Ophthalmic Solution (OS) 2% Versus Timoptol® XE Ophthalmic Solution (OS) 0.5% in Ocular Hypertension Patients
Brief Title: A Study to Evaluate Efficacy and Safety Effects Using Mikelan® LA Ophthalmic Solution (OS) 2% Versus Timoptol® XE Ophthalmic Solution (OS) 0.5% in Ocular Hypertension Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Taiwan Otsuka Pharm. Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 001-TWB-0901(n)
Record Dates: First submitted 2009-08-20; First posted 2009-09-07 (Estimated); Last update posted 2011-09-05 (Estimated); Status verified 2011-09

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — Carteolol; Timolol; Latanoprost

ARMS (2):
- Treatment A Group (Experimental): Mikelan LA + Xalatan
  Interventions: Drug: carteolol (Mikelan), timolol (Timoptol), latanoprost (Xalatan)
- Treatment B Group (Active Comparator): Timoptol XE + Xalatan
  Interventions: Drug: carteolol (Mikelan), timolol (Timoptol), latanoprost (Xalatan)

INTERVENTIONS:
Drug: carteolol (Mikelan), timolol (Timoptol), latanoprost (Xalatan) — Experimental: Mikelan, 1 drop/daily, for 8 weeks Active Comparator: Timoptol, 1 drop/daily, for 8 weeks

SUMMARY:
The primary objective of the clinical study is to evaluate the efficacy and safety for Mikelan LA eye drops 2% (once per day) of intra-ocular pressure decreased.

ELIGIBILITY:
Inclusion Criteria:

1. Male or females outpatients with primary open-angle glaucoma or ocular hypertension;
2. Subjects who have received Latanoprost at least 4 weeks, and in the end of screening period, subject's Intra-Ocular Pressure is ≧18mmHg (choice of one eyes is possible), or Investigator judges the reduction of IOP is insufficient of individual subject.
3. Aged between ≧ 20 and ≦80 years old when giving informed consent to the study.

Exclusion Criteria:

1. Hypersensitivity to either oral or topical beta-blocker therapy or to any ophthalmic solution used in the study;
2. Patients wearing contact lenses;
3. Patients with severe dry eyes;
4. Patients who had ophthalmic surgery including cataract surgery, trabeculotomy or trabeculectomy within three months of study start;
5. Patients who had laser trabeculoplasty within 2 months before starting study;
6. Patients who had corneal contamination, and acute ophthalmic infection, or inflammatory ophthalmic disorder 2 months before starting study;
7. Patients who had herpetic keratitis or corneal ulcer within 2 months before starting study;
8. Patient who are receiving systemic administration of drugs that may have and effect on IOP;
9. Patients who have poorly controlled heart failure, sinus bradycardia, atrioventricular block (1 and 2 grade), or cardiogenic shock;
10. Patients with brochial asthma, bronchospasm or severe chronic obstructive pulmonary disease or a history thereof;
11. Patients with poorly controlled diabetes or diabetic ketoacidosis or metabolic acidosis;
12. Patients with aortic stenosis, Raynaud's syndrome, intermittent claudication, or pheochromocytoma;
13. Patients with myasthenia gravis;
14. Patients with severe hepatic or renal disorder judged by investigator;
15. Patients who have confirmed or potential pregnancy, current lactation, or wish to become pregnant during the study period;
16. Patients who have treatment with any investigational drug when giving informed consent;
17. Patients with significant alcohol, drug or medication abuse as judged by investigator;
18. Patients whom investigator judges as subjects to be inappropriate for the clinical study (e.g., patient with severe complication)

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2009-10; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
The change value of Intra-Ocular Pressure (IOP) in study group | assessment will be done every month for 2 months for each subject

SECONDARY OUTCOMES:
The change value of IOP between groups | assessment will be done every month for 2 months for each subject
The change percentage of IOP in each group | assessment will be done every month for 2 months for each subject
The change of score of Patient satisfaction in each group | assessment will be done every month for 2 months for each subject

CONTACTS AND LOCATIONS:
Overall Officials: Da-Wen Lu, MD/PhD, Principal Investigator — Department of Opthalmology/ Tri-Service General Hospital
Locations (1):
- Tri-Service General Hospital, Taipei, Taiwan